CLINICAL TRIAL: NCT03032094
Title: Connective Tissue Grafting for Single Tooth Recession Defects & the Impact of the Thickness of the Palatal Harvest Tissue: A Pilot Study
Brief Title: Connective Tissue Grafting for Single Tooth Recession & the Impact of the Thickness of the Palatal Harvest Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Evanthia Lalla, Professor of Dental Medicine (Periodontics), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAN2667
Record Dates: First submitted 2017-01-11; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Gingival Recession
Keywords: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1mm thick graft (Active Comparator): connective tissue graft of 1mm thickness
  Interventions: Procedure: connective tissue graft
- 2mm thick graft (Active Comparator): connective tissue graft of 2mm thickness
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Procedure: connective tissue graft — palatal connective tissue graft to attain root coverage

SUMMARY:
The purpose of this study is to test if the thickness of the graft taken from the roof of the mouth, has a significant effect on the amount of attached tissue and the amount of root coverage that are attained when treating a single tooth with gingival recession.

DETAILED DESCRIPTION:
The goal of the study is to determine if the thickness of a tissue graft taken from the roof of the mouth, used to cover the exposed root of a tooth, affects the overall outcome of the root coverage, the health of the resulting tissue, as well as postoperative pain as reported by the patient. Connective tissue grafts will be harvested in different thicknesses, and results of the procedures will be compared. Qualified subjects will undergo a root coverage procedure, after random assignment to one of the groups. Regular recall visits to monitor healing at intervals of 1 week, 2 weeks, 1 month, and 3 months will be scheduled. Subjects will be asked to fill out patient response forms regarding pain and other symptoms at these visits. Photographs will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old
2. Absence of active periodontal disease
3. Single tooth (premolars and anterior teeth) with Miller class I or II gingival recession >= 2mm
4. Detectable Cemento-Enamel Junction (CEJ) -

Exclusion Criteria:

1. Smokers (>10 cigarettes/ per day)
2. Uncontrolled systemic diseases with compromised healing potential (DM with HbA1c >7%)
3. Active infectious diseases (hepatitis, tuberculosis, HIV, etc.)
4. Medication known to cause gingival enlargement
5. Patients taking anticoagulants with an international normalized ratio (INR) >2.5
6. Long-term (>2 weeks) use of antibiotics in the past 3 months
7. Pregnant or attempting to get pregnant
8. Sites with probing depth > 4mm
9. Recession adjacent to an edentulous area
10. Frenal and muscle attachment that encroach on the marginal gingiva

    a. Can be included 2 months after surgical therapy to remove the frenum (frenectomy)
11. History of periodontal surgical treatment of the involved sites
12. Prosthetic crown, restorations or caries in the candidate tooth and adjacent teeth
13. Teeth with pulpal pathology
14. Severe teeth malposition and open contacts
15. Planned orthodontic treatment to commence within 1 year following procedure
16. Parafunctional habits -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Root coverage | Upto 3 months
  Amount of root coverage attained in millimeters
Root coverage | Upto 3 months
  Amount of root coverage attained in percentage
width of keratinized tissue | Upto 3 months
  Amount of zone of keratinized tissue attained in millimeters
width of keratinized tissue | Upto 3 months
  Amount of zone of keratinized tissue attained in percentage

SECONDARY OUTCOMES:
thickness of keratinized tissue | Upto 3 months
amount of erythema and edema | Upto 3 months
  patient reported outcome of amount of erythema and edema in number of days postoperatively
duration of erythema and edema | Upto 3 months
  patient reported outcome of duration of erythema and edema in number of days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Lalla, DDS, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided